CLINICAL TRIAL: NCT04067544
Title: Acupuncture Treatment of Chemotherapy-Induced Peripheral Neuropathy in Women With Breast or Gynecologic Cancers: Mechanisms of Action and Feasibility
Brief Title: Acupuncture Treatment of Chemotherapy-Induced Peripheral Neuropathy in Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unforeseen complications due to COVID-19 and funding
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 107709
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2023-11

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Breast Cancer Female; Gynecologic Cancer
Keywords: paclitaxel; chemotherapy-induced peripheral neuropathy; breast cancer; gynecologic cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Acupuncture Treatment (Experimental): All participants receive 10 acupuncture treatments over the course of 8 weeks.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — The manualized acupuncture treatment (AT) intervention will be designed by Dr. Budhathoki and Dr. Taylor-Swanson and administered by Dr. Budhathoki and members of Huntsman acupuncture team. Ten sessions of AT will be delivered: twice per week for 2 weeks, thereafter once per week for six weeks, with a total of 9 treatments during a two-month course. Each session will last 45-60 minutes, with acupuncture needles retained 30-40 minutes. A minimum of 8 treatments must be received by each participant with no more than 9 days' gap between treatments permitted. Concurrent medications are allowed as prescribed and will be tracked in the study and analyzed as potential confounders.
  Participants in the study will undergo study interview and fMRI at the following two time points: within 9 days after baseline following enrollment and within one week of acupuncture treatment completion.

SUMMARY:
This pilot study aims to evaluate the feasibility to conduct a study of acupuncture treatment (AT) for Chemotherapy-Induced Peripheral Neuropathy (CIPN) at Huntsman Cancer Institute and to investigate changes in physiological biomarkers when using acupuncture to treat CIPN.

DETAILED DESCRIPTION:
This pilot feasibility study aims to determine if conducting a trial of AT for CIPN is feasible at Huntsman Cancer Institute (HCI). The investigators aim to enroll and retain twenty participants who will undergo fMRI during the baseline visit, receive 10 sessions of AT, and undergo fMRI after completion of AT. The investigators will examine fMRI for potential neurologic mechanisms of action of AT in CIPN management. The ultimate objective of this pilot project is to lay the foundation for a future randomized controlled clinical trial of AT for CIPN. Specifically, the investigators will be able to demonstrate that the investigators have the team and location in place to conduct a successful trial.

The participant will receive 10 acupuncture treatments over the course of 8 weeks with a baseline fMRI done prior to receiving acupuncture treatments and a final fMRI done after the completion of acupuncture treatments. Participant will receive questionnaires before fMRI, acupuncture treatments following final fMRI and at a 3 month follow up time point. (See below for more detail.)

1.1 Primary Objectives and Endpoints

To evaluate the feasibility to conduct a trial of AT for CIPN + standard of care therapy. Primary feasibility objectives will be evaluated in terms of recruitment (enrollment of 20 women, average of 2 eligible women per month to participate in the trial, identification of appropriate recruitment strategies, the appropriateness of eligibility criteria), retention (70% or more participants comply with 8 or more AT sessions and complete both fMRI scans), safety (zero serious adverse events directly related to AT) and questionnaire completion (70% or more enrolled participants comply with all data collection).

1.1.1 Primary outcome measures: Mean enrollment, completion rate of AT, fMRI, rate of serious adverse events, rate of questionnaire completion.

1.2 Secondary Objectives and Endpoints To evaluate the impact of AT on the reported experience of CIPN. 1.2.1 To evaluate central pain processing and cortical connectivity in patients with CIPN treated by acupuncture by analyzing fMRI of all participants.

1.2.2 To evaluate if there is any change in patient-reported measures from before AT to after study completion.

This study will enroll female patients who have completed treatment with paclitaxel or docetaxel at least three months prior. Paclitaxel and docetaxel are neurotoxic chemotherapies known to cause CIPN. Patients must have experienced at least one month of altered sensation and/or pain with a score of greater than or equal to 20 for CIPN on the sensory subscale of the CIPN-20. The investigators will commence recruitment 3 months after patients have completed their last paclitaxel or docetaxel dose. Patients will be recruited from the Huntsman Cancer Center Oncology Clinics in collaboration with their oncologists.

For this study, enrollment will be limited to patients with breast, ovarian, cervical, endometrial, or uterine cancer with CIPN and completed paclitaxel or docetaxel treatments.

Visits:

Screening Visit:

Potentially eligible subjects will be scheduled for a screening visit. After informed consent is obtained, the Study Coordinator (SC) will review and confirm inclusion/exclusion criteria. The SC will take a brief medical and neurological history and administer the CIPN-20 questionnaire. If all inclusion and exclusion criteria are fulfilled, the subject will proceed to baseline visit. This visit may occur on the same day as screening, but must occur within 2 weeks of study screening visit.

Baseline Visit:

Patients diagnosed with breast, ovarian, cervical, endometrial, or uterine cancer who were treated with paclitaxel or docetaxel chemotherapy associated with CIPN will undergo a number of questionnaires/exam scales designed to assess neuropathic symptoms and the effect of neuropathy on quality of life. The patient will then be enrolled in the study and scheduled in the Wellness Center for acupuncture therapy (AT). All participants will be scheduled for fMRI , which must occur within nine days after baseline.

Participants will undergo study interview and fMRI within 9 days after baseline following enrollment.

Demographic data and clinical data including current medications and medical history and fall rates will be gathered during the baseline visit. Questionnaires (BPI, CIPN-20, CIPN- Rasch-built Overall Disability Scale (R-ODS), MAIA-2) will be completed in person or emailed to patients via REDCap at baseline. Reminder calls and AT appointments will be scheduled by HCI Wellness and Integrative Health Center personnel in conjunction with a SC. The SC will aid participants in scheduling fMRI appointments online. AT treatments will occur within 7 days/4 business days in general.

Follow up Visits:

Participants will receive 10 sessions of AT: twice per week for 2 weeks, thereafter once per week for six weeks, with a total of 10 treatments during a two-month course. Each session will last 45-60 minutes, with acupuncture needles retained 30-40 minutes. A minimum of 8 treatments must be received by each participant with no more than 9 days' gap between weekly treatments permitted (sessions 5-10). Concurrent medications are allowed as prescribed and will be tracked in the study and analyzed as potential confounders.

Final Visit:

Participants will undergo examination within one week of AT completion. This will include the fMRI scan and questionnaires. Compensation for participation will be offered following the completion of questionnaires.

Measures:

Questionnaires will be completed in person or emailed to patients via REDCap at baseline and study conclusion, as well as at a 3-month follow-up. Primary Endpoints: Mean enrollment, percentage completion rate of all study procedures, frequency count of serious adverse events, and percentage of enrolled participants completing questionnaires will be calculated. Data will be collected via REDCap and analyzed with Statistical Package for the Social Sciences (SPSS).

Additional measures to be collected: CIPN-20: This measure includes questions about tingling, numbness, painful numbness, cramps, balance, temperature intolerance, grasping items, ankle flexion weakness and leg weakness. CIPN-R-ODS (a validated measure of quality of life specific to CIPN), will be used to assess impact on function, BPI to assess pain and Multidimensional Assessment of Interoceptive Awareness (MAIA-2) to assess mind-body awareness. The investigators will also collect demographic information including age, marital status, race and ethnicity, current medications and medical history.

Acupuncture therapy (AT): AT will be delivered onsite at HCI in the Linda B. and Robert B. Wiggins Wellness & Integrative Health Center. AT will be delivered twice per week for two weeks and then weekly for six weeks by Annie Budhathoki, Doctor of Acupuncture and Oriental Medicine (DAOM), a Licensed Acupuncturist who has over five years' clinical experience treating persons with cancer, or another Licensed Acupuncturist in the Wellness & Integrative Health Center. Each session will last 45-60 minutes, with acupuncture needles retained 30-40 minutes. A minimum of 8 treatments must be received by each participant with no more than 9 days' gap between weekly treatments permitted (sessions 5-10). .

Functional MRI (fMRI) to be conducted within 9 days after baseline and within 1 week of final AT session. fMRI scans will be conducted at Imaging and Neuroscience Center (INC) in Research Park. Imaging will consist of structural brain imaging (MP2RAGE), task fMRI, and resting-state fMRI connectivity. Task fMRI will consist of a mental imagery task with a 20-second block design wherein patients will alternate between concentration on a part of their body where they experience pain and a part of their body where they do not experience pain, prompted by visual cues. The investigators will provide gift cards for $25 after the completion of the second fMRI and questionnaires associated with this visit.

Clinical evaluations: Demographic data, clinical data including current medications and medical history and fall rates will be gathered.

ELIGIBILITY:
Inclusion Criteria:

Female age 18 or older.

* Histologically proven breast, uterine, cervical or ovarian cancer of any stage.
* Received either (1) a Paclitaxel treatment dose of at least 480 mg/m2 paclitaxel as a single or combination agent or (2) a Docetaxel treatment dose of at least 150 mg/m2 docetaxel as a single or combination agent. Treatment must be completed at least 3 months prior to enrollment.
* Eligible participants report at least 1 month of altered sensation and/or pain in the feet (with or without presence in one or both hands) with a score of greater than or equal to 20 for CIPN on the sensory subscale of the CIPN-20 (scale 0-100).
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Eastern Cooperative Oncology Group (ECOG) status of 0 (asymptomatic), 1 (symptomatic but completely ambulatory) or 2 (symptomatic, <50% in bed during the day).

Exclusion Criteria:

* Preexisting neuropathy due to other identified etiologies includes diabetes, vitamin B12 deficiency, or alcoholism.
* Having received more than 6 acupuncture treatments for any condition in the last six months.
* Participants with claustrophobia, pacemakers, non-MRI compatible breast expanders or port-a-caths, neurostimulator devices, current pregnancy, exposure to shrapnel, left-handedness, or otherwise unsafe for MRI scanning.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Taylor-Swanson, PhD LAc, Principal Investigator — Associate Professor of College of Nursing, Licensed Acupunturist
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture Treatment: All participants receive 10 acupuncture treatments over the course of 8 weeks.
  Acupuncture: The manualized acupuncture treatment (AT) intervention will be designed by Dr. Budhathoki and Dr. Taylor-Swanson and administered by Dr. Budhathoki and members of Huntsman acupuncture team. Ten sessions of AT will be delivered: twice per week for 2 weeks, thereafter once per week for six weeks, with a total of 9 treatments during a two-month course. Each session will last 45-60 minutes, with acupuncture needles retained 30-40 minutes. A minimum of 8 treatments must be received by each participant with no more than 9 days' gap between treatments permitted. Concurrent medications are allowed as prescribed and will be tracked in the study and analyzed as potential confounders.
  Participants in the study will undergo study interview and functional magnetic resonance imaging (fMRI) at the following two time points: within 9 days after baseline following enrollment and within one week of acupuncture treatment completion.
Period: Overall Study
Arm/Group | Acupuncture Treatment
Started | 3
Completed | 2
Not Completed | 1
Not completed — Unforeseen recruitment issues due to Coronavirus Disease (COVID)-19 pandemic | 1

BASELINE CHARACTERISTICS:
Groups:
- Acupuncture Treatment: All participants receive 10 acupuncture treatments over the course of 8 weeks.
  Acupuncture: The manualized acupuncture treatment (AT) intervention will be designed by Dr. Budhathoki and Dr. Taylor-Swanson and administered by Dr. Budhathoki and members of Huntsman acupuncture team. Ten sessions of AT will be delivered: twice per week for 2 weeks, thereafter once per week for six weeks, with a total of 9 treatments during a two-month course. Each session will last 45-60 minutes, with acupuncture needles retained 30-40 minutes. A minimum of 8 treatments must be received by each participant with no more than 9 days' gap between treatments permitted. Concurrent medications are allowed as prescribed and will be tracked in the study and analyzed as potential confounders.
  Participants in the study will undergo study interview and fMRI at the following two time points: within 9 days after baseline following enrollment and within one week of acupuncture treatment completion.
Arm/Group | Acupuncture Treatment
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Participant reported symptoms at baseline [Mean (Standard Deviation); unit: score on a scale] — The 20-item questionnaire is scored using a four-point Likert-type scale ranging from 1 (not at all) to 4 (very much), and evaluates sensory (9 items), motor (8 items), and autonomic (3 items for men, 2 items for women) symptom subscales. Items from each subscale are summed, then linearly converted to a 0-100 scale. The three subscale scores are averaged to obtain a total score, with the final score range being 0-100. For raw and scaled scores, higher scores indicate more symptoms of peripheral neuropathy. Only participants who completed all questionnaires were included. Population: Only participants who completed all questionnaires were evaluable for the questionnaire-related outcome (i.e. Outcome 6), so this baseline measure also only reports questionnaires completed by participants who were evaluated for that outcome.
  score on a scale
    number analyzed (Participants) | 2
    (all) | 74.13 (15.468)

OUTCOME MEASURES:

1. Primary Outcome: Mean Monthly Enrollment
Description: We calculated the mean number of participants who enrolled per month while the study was open to accrual.
Time Frame: 7 Months
Measure: Mean (Standard Deviation); unit: participants per month
Arm/Group | Acupuncture Treatment
Number analyzed (Participants) | 3
participants per month | 0.429 (0.787)

2. Primary Outcome: Number of Participants Compliant With Treatment
Description: Participant retention was defined as the number of participants who attended at least 8 out of 10 AT sessions and completed both fMRI scans
Time Frame: 7 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture Treatment
Number analyzed (Participants) | 3
Participants | 2

3. Primary Outcome: Number of Participants Who Experience Serious Adverse Events Related to AT Sessions
Description: A serious adverse event is any undesirable experience associated with the participation in this study in a participant that results in death, life-threatening conditions, hospitalization, disability or permanent damage or birth defect.
Time Frame: 7 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture Treatment
Number analyzed (Participants) | 3
Participants | 0

4. Primary Outcome: Number of Participants Who Completed Questionnaires
Description: Participants who completed all questionnaires, which were administered at baseline and at 3 months post-treatment.
Time Frame: 7 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture Treatment
Number analyzed (Participants) | 3
Participants | 2

5. Secondary Outcome: Change in Functional Connectivity of Central Pain Networks on fMRI (Z-scores)
Description: Connectivity changes were evaluated using resting-state fMRI at baseline and post-treatment. Independent component analysis was used to identify networks, and statistical thresholds were applied to define significant changes. Z-scores represent standard deviations from the mean of a normative reference population, with positive values indicating increased connectivity and negative values indicating decreased connectivity.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Acupuncture Treatment
Number analyzed (Participants) | 2
Z-Score | 3.32 (0.59)

6. Secondary Outcome: Change in Participant-reported Symptoms From Before AT to After Study Completion
Description: Quality of Life Questionnaire (QLQ) - Chemotherapy Induced Peripheral Neuropathy (CIPN) 20 (QLQ-CIPN-20) questionnaire is administered to participants at baseline (BL) and at 3 months post-treatment (approximately 22 weeks total between time points). Mean difference between BL and 3 Month Questionnaire scores will be calculated. Only participants who have completed all questionnaires will be evaluated. The 20-item questionnaire is scored using a four-point Likert-type scale ranging from 1 (not at all) to 4 (very much), and evaluates sensory (9 items), motor (8 items), and autonomic (3 items for men, 2 items for women) symptom subscales. Items from each subscale are summed, then linearly converted to a 0-100 scale. The three subscale scores are averaged to obtain a total score, with the final score range being 0-100. For raw and scaled scores, higher scores indicate more symptoms of peripheral neuropathy.
Time Frame: 22 weeks
Population: Only 2 participants completed all 3 questionnaires so only these scores were used.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Acupuncture Treatment
Number analyzed (Participants) | 2
change in score on a scale | -25.17 (5.156)

7. Other Pre Specified Outcome: Participant Reported Symptoms 3 Months Post Treatment
Description: Quality of Life Questionnaire-Chemotherapy Induced Peripheral Neuropathy 20 (QLQ-CIPN-20) questionnaire is administered to participants at baseline (BL) and at 3 months post-treatment (approximately 22 weeks total between time points). This outcome reports mean participant scores at 3 months post treatment. Only participants who have completed all questionnaires will be evaluated. The 20-item questionnaire is scored using a four-point Likert-type scale ranging from 1 (not at all) to 4 (very much), and evaluates sensory (9 items), motor (8 items), and autonomic (3 items for men, 2 items for women) symptom subscales. Items from each subscale are summed, then linearly converted to a 0-100 scale. The three subscale scores are averaged to obtain a total score, with the final score range being 0-100. For raw and scaled scores, higher scores indicate more symptoms of peripheral neuropathy.
Time Frame: 22 weeks
Population: Only two participants completed questionnaires at 3 months post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture Treatment
Number analyzed (Participants) | 2
score on a scale | 48.96 (20.624)

ADVERSE EVENTS:
Time Frame: From start of acupuncture treatment (AT) to 12 weeks following discontinuation of AT (approximately 22 weeks per patient)
Arm/Group | Acupuncture Treatment
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupuncture Treatment (N=3)
localized edema (General disorders) | 1 (1) — Arm swelling
Nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic forced recruitment and enrollment to stop in March 2020 leading to small numbers of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT04067544/Prot_SAP_000.pdf